CLINICAL TRIAL: NCT02746952
Title: Phase I, Open Label, Dose-escalation Study Followed by a Safety Expansion Part to Evaluate the Safety, Expansion and Persistence of a Single Dose of UCART19 (Allogeneic Engineered T-cells Expressing Anti-CD19 Chimeric Antigen Receptor), Administered Intravenously in Patients With Relapsed or Refractory CD19 Positive B-cell Acute Lymphoblastic Leukaemia (B-ALL)
Brief Title: Dose Escalation Study of UCART19 in Adult Patients With Relapsed / Refractory B-cell Acute Lymphoblastic Leukaemia
Acronym: CALM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-68587-002; 2016-000296-24 (EudraCT Number)
Record Dates: First submitted 2016-03-07; First posted 2016-04-21 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UCART19 (Experimental)
  Interventions: Biological: UCART19

INTERVENTIONS:
Biological: UCART19
  Other Names: S68587

SUMMARY:
The study is in two parts: a dose escalation then a safety dose expansion. The purpose of the dose escalation part is to evaluate the safety and tolerability of ascending doses of UCART19 (dose-escalation part) given as a single infusion in patients with relapsed / refractory (R/R) B-cell acute lymphoblastic leukaemia (B-ALL), to determine the maximum tolerated dose (MTD), the recommended dose and the lymphodepletion regimen. The purpose of the safety dose expansion is to assess the safety and tolerability of the RD for UCART19.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant
* Age ≥ 16 years
* Patient with relapsed or refractory CD19 positive B-acute lymphoblastic leukaemia (B-ALL) who have exhausted alternative treatment options
* Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
* Eastern Cooperative Oncology Group (ECOG) performance status < 2

Exclusion Criteria:

* Previous treatment with gene or gene-modified cell therapy medicine products or adoptive T cell therapy
* Use of previous anti-leukemic therapy (including approved therapies and other investigational products) within 5 half-lives prior to UCART19 administration
* CD19 negative B-cell leukaemia
* Burkitt cell or mixed lineage acute leukaemia

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Dose escalation part: Dose Limiting Toxicities (DLTs) occurence. Dose expansion part: AE throughout the study. | Dose Escalation: Up to day 28 post first UCART19 infusion. Dose Expansion: From inclusion to Month 12

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | From inclusion to Month 12
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Objective Remission Rate | At Day 28, Day 84, Month 4, Month 6, Month 9 and Month12
  Proportion of patients in whom a response among molecular complete remission (mCR), morphologic complete remission (CR) and complete remission with incomplete blood count recovery (CRi)
Duration of remission | From the time that response criteria are first met until the date of progression or death (whatever the reason of death), whichever occurs first, assessed up to Month 12
Time to remission | From the date of UCART19 administration until the date that response criteria are met, assessed up to Month 12
Progression Free Survival (PFS) | From the date of UCART19 administration until the date of progression or the date of death (whatever the reason of death), whichever occur first, assessed up to Month 12
Overall Survival (OS) | From the date of UCART19 administration to the date of death from any cause, assessed up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Benjamin, MD, PhD, Principal Investigator — King's College Hospital NHS Trust
Locations (9):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
- Japan (2):
  - Kyushyu University Hospital, Fukuoka
  - Hokkaido University Hospital, Sapporo
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Result] Benjamin R, Graham C, Yallop D, Jozwik A, Mirci-Danicar OC, Lucchini G, Pinner D, Jain N, Kantarjian H, Boissel N, Maus MV, Frigault MJ, Baruchel A, Mohty M, Gianella-Borradori A, Binlich F, Balandraud S, Vitry F, Thomas E, Philippe A, Fouliard S, Dupouy S, Marchiq I, Almena-Carrasco M, Ferry N, Arnould S, Konto C, Veys P, Qasim W; UCART19 Group. Genome-edited, donor-derived allogeneic anti-CD19 chimeric antigen receptor T cells in paediatric and adult B-cell acute lymphoblastic leukaemia: results of two phase 1 studies. Lancet. 2020 Dec 12;396(10266):1885-1894. doi: 10.1016/S0140-6736(20)32334-5. PMID 33308471
- [Derived] Benjamin R, Jain N, Maus MV, Boissel N, Graham C, Jozwik A, Yallop D, Konopleva M, Frigault MJ, Teshima T, Kato K, Boucaud F, Balandraud S, Gianella-Borradori A, Binlich F, Marchiq I, Dupouy S, Almena-Carrasco M, Pannaux M, Fouliard S, Brissot E, Mohty M; CALM Study Group. UCART19, a first-in-class allogeneic anti-CD19 chimeric antigen receptor T-cell therapy for adults with relapsed or refractory B-cell acute lymphoblastic leukaemia (CALM): a phase 1, dose-escalation trial. Lancet Haematol. 2022 Nov;9(11):e833-e843. doi: 10.1016/S2352-3026(22)00245-9. Epub 2022 Oct 10. PMID 36228643
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/